CLINICAL TRIAL: NCT06714175
Title: Effects of Lower Limb Leg Press Power Training Combined with Visual Feedback Games on Physical Performance, Cognitive Function, and Heart Rate Variability in the Elderly
Brief Title: Leg Press Power Training with Visual Feedback Games Improves Physical, Cognitive, and Heart Health in Seniors
Acronym: LPPT-VFG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Yi-Wei Kao, Principal Investigator, Kaohsiung Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-202 20046; KMUHIRB-F(II)-202 20046 (Other: Kaohsiung Medical University Chung-Ho Memorial Hospital Institutional Review Board)
Record Dates: First submitted 2024-11-13; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Elderly (people Aged 65 or More)
Keywords: Elderly; Muscle Strength; Lower Limb Power Training; Visual Feedback Games; Cognitive Function; Heart Rate Variability; Resistance Training
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with a parallel assignment model. Participants are randomly assigned to either the experimental group or the control group. The experimental group undergoes lower limb leg press power training combined with visual feedback games twice a week for 12 weeks, while the control group maintains their usual daily activities. The outcomes are assessed before and after the 12-week intervention, focusing on physical performance, cognitive function, and heart rate variability (HRV).
Masking Description: Two long-term care centers were selected for the study. One center was randomly assigned to the experimental group through a lottery system, while the other served as the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): This group will not receive any specific muscle power intervention.
- Lower Limb Strength Training Program with Visual Feedback (Experimental): This lower limb explosive strength training system integrates visual feedback games and is equipped with angle and force sensors to simultaneously output the power of the left and right legs, as well as maximum explosive force and pushing force. Users can immediately understand the balance of leg strength and make adjustments, making it particularly suitable for the elderly to improve lower limb strength or for rehabilitation training. The gamification of the system enhances the fun of training, while data quantification allows progress tracking, making the training more precise and effective. Additionally, after the game ends, data can be exported to Excel for further analysis to identify issues in the pushing process and optimize the training plan.
  Interventions: Behavioral: Lower Limb Strength Training Program with Visual Feedback

INTERVENTIONS:
Behavioral: Lower Limb Strength Training Program with Visual Feedback — This lower limb explosive strength training system integrates visual feedback games and is equipped with angle and force sensors to simultaneously output the power of the left and right legs, as well as maximum explosive force and pushing force. Users can immediately understand the balance of leg strength and make adjustments, making it particularly suitable for the elderly to improve lower limb strength or for rehabilitation training. The gamification of the system enhances the fun of training, while data quantification allows progress tracking, making the training more precise and effective. Additionally, after the game ends, data can be exported to Excel for further analysis to identify issues in the pushing process and optimize the training plan.
  Arms: Lower Limb Strength Training Program with Visual Feedback

SUMMARY:
This study investigates the effects of lower limb leg press power training combined with visual feedback games on the physical performance, cognitive function, and heart rate variability (HRV) of older adults aged 65 and above. Participants were divided into an experimental group and a control group, with the experimental group engaging in leg press exercises combined with visual games twice a week for 12 weeks.

DETAILED DESCRIPTION:
This study aims to investigate the effects of lower limb leg press power training combined with visual feedback games on the physical and cognitive health of the elderly. With the aging population increasing, the decline in muscle strength and cognitive function has become a significant challenge for older adults. To address these health issues, this study plans to recruit 40 participants aged 65 and above and randomly assign long-term care centers into an experimental group and a control group. The experimental group will perform leg press training combined with visual feedback games twice a week for 12 weeks, while the control group will continue their usual daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years old
* Physical fitness and health assessment results are suitable for exercise
* Clear consciousness and no mental disorders .
* Able to walk independently for more than 10 meters.

Exclusion Criteria:

* Determined by doctors or other relevant professionals that they cannot accept cardiopulmonary testing and muscle strength training
* The resting heartbeat exceeds 120 beats per minute, the systolic blood pressure exceeds 160mmHg, and the diastolic blood pressure exceeds 100mmHg.
* Any stage of cancer and other hematologic diseases that affect research evaluation, such as: severe anemia.
* Diseases related to cardiac pacemakers and arrhythmias.
* Other neurological, muscular, or skeletal diseases that may affect the research assessment or severe contagious disease.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Testing will be conducted in Week 0, Week 6, and Week 13
  Measurement of lower limb muscle strength (pound), including the quadriceps and hamstrings
Muscle Strength | Testing will be conducted in Week 0, Week 6, and Week 13
  hand grip strength (kilogram)

SECONDARY OUTCOMES:
Physiological Data | Testing will be conducted in Week 0, Week 6, and Week 13.
  Height (centimeters)
Physiological Data | Testing will be conducted in Week 0, Week 6, and Week 13
  weight (kilogram)
Physiological Data | Testing will be conducted in Week 0, Week 6, and Week 13
  systolic and diastolic blood pressure (mmHg)
Physiological Data | Testing will be conducted in Week 0, Week 6, and Week 13
  blood oxygen (SaO2)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  AVG HR (average heart rate)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  HRV (heart rate variability)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  RMSSD (root mean square of successive differences)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  SDNN (standard deviation of NN intervals)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  M RR int. (mean RR interval)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13.
  TP (total power)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13
  LF (low frequency power in ms² and Hz)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13
  HF (high frequency power in ms² and Hz)
Heart Rate Variability (HRV) | Baseline measurement at Week 0 and follow-up measurement at Week 13
  LF/HF ratio
Cognitive Function Assessment | Baseline measurement at Week 0 and follow-up measurement at Week 13
  Cognitive function is assessed using the Taiwan Chinese version of the Montreal Cognitive Assessment (MoCA), authorized by the original Korean publisher. This assessment evaluates various cognitive domains to provide a comprehensive understanding of cognitive health.
Physical Performance Assessment | Testing will be conducted in Week 0, Week 6, and Week 13
  Physical performance is evaluated using the Short Physical Performance Battery (SPPB)
Physical Performance Assessment | Testing will be conducted in Week 0, Week 6, and Week 13
  The 30-Second Sit-to-Stand Test
Physical Performance Assessment | Baseline measurement at Week 0 and follow-up measurement at Week 13
  Functional Reach Test

CONTACTS AND LOCATIONS:
Overall Officials: GUO L Y Professor and Dean of the College of Health Sciences, Departme, Ph.D., Study Chair — Department of Sports Science, Kaohsiung Medical University, Taiwan
Locations (1):
- Lower Limb Power Training Exercise Equipment, Kaohsiung City, Taiwan, No. 100, Shiquan 1st Road, Sanmin District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
This study aims to investigate the effects of lower limb leg press power training combined with visual feedback games on the physical and cognitive health of the elderly. With the aging population increasing, the decline in muscle strength and cognitive function has become a significant challenge for older adults. To address these health issues, this study plans to recruit 40 participants aged 65 and above and randomly assign long-term care centers into an experimental group and a control group. The experimental group will perform leg press training combined with visual feedback games twice a week for 12 weeks, while the control group will continue their usual daily activities.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting information will be available starting 2 years after the publication of the primary study results and will remain accessible for 5 years.
Access Criteria: The related supporting documents will only be made available to qualified researchers affiliated with academic institutions, medical organizations, or public health agencies. Applicants must submit a detailed research proposal and ethical approval documents, and access will be granted only upon approval.